CLINICAL TRIAL: NCT01695369
Title: Clinical Comfort Evaluation of Biofinity and Acuvue Oasys Lenses
Brief Title: Evaluation of Comfilcon A and Senofilcon A Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: CV-12-54
Record Dates: First submitted 2012-09-26; First posted 2012-09-28 (Estimated); Results first posted 2014-03-06 (Estimated); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Senofilcon A (Active Comparator): Senofilcon A; Comfilcon A
  Interventions: Device: Senofilcon A; Comfilcon A; Device: Comfilcon A; Senofilcon A
- Comfilcon A (Experimental): Comfilcon A; Senofilcon A
  Interventions: Device: Senofilcon A; Comfilcon A; Device: Comfilcon A; Senofilcon A

INTERVENTIONS:
Device: Senofilcon A; Comfilcon A — Senofilcon A; Comfilcon A
Device: Comfilcon A; Senofilcon A — Comfilcon A; Senofilcon A

SUMMARY:
Evaluation of Comfilcon A and Senofilcon A Lenses

DETAILED DESCRIPTION:
Non-dispensing, single-masked, randomized, contralateral study comparing the test lens against the control lens. Each subject will be randomized to wear the test lens in one eye and the control lens in the other eye.

ELIGIBILITY:
Inclusion Criteria:

Subjects must satisfy the following conditions prior to inclusion in the study:

* Has had an oculo-visual examination in the last two years
* Is at least 18 years of age and has full legal capacity to volunteer
* Has read and understood the information consent letter
* Is willing and able to follow instructions and maintain the appointment schedule
* Is correctable to a visual acuity of 20/30 or better (in each eye) with their habitual vision correction
* Currently wears soft contact lenses at least 3 days a week, 8 hours a day
* Has clear corneas and no active ocular disease
* Has not worn lenses for at least 12 hours before the examination
* Have normal eyes with no evidence of abnormality or disease. For the purposes of this study a normal eye is defined as one having:

  * No amblyopia
  * No evidence of lid abnormality or infection (e.g. entropion, ectropion, chalazia, recurrent styes)
  * No clinically significant slit lamp findings (e.g. infiltrates or other slit lamp findings Grade 2 or above: corneal edema, tarsal abnormalities, and conjunctival injection).
  * No other active ocular disease (e.g. glaucoma, history of recurrent corneal erosions, cornea [infiltrates], conjunctiva, lids, and intraocular infection or inflammation of an allergic, bacterial, or viral etiology)
  * No aphakia
  * Has prescription to match the available power range.

Exclusion Criteria:

Any of the following will render a subject ineligible for inclusion:

* Greater than 0.75 of refractive astigmatism in either eye
* Has never worn contact lenses before
* Wears contact lenses on an extended wear basis
* Has any systemic disease affecting ocular health
* Is a known sufferer of ocular allergies
* Is taking medication, such as oral antihistamines, antihistamine eye drops, oral and ophthalmic beta-adrenergic blockers (e.g. Propanolol, Timolol), anticholinergics, oral steroids and any prescribed or over-the-counter eye medication, except artificial tears or eye lubricants
* Has any clinically significant lid or conjunctival abnormalities, neovascularization, corneal scars or corneal opacities
* Is aphakic
* Has undergone corneal refractive surgery.
* Is wearing monovision
* Is participating in any other type of clinical or research study
* Female who is currently pregnant or is breast-feeding
* Has > grade 1 ocular corneal staining in both type and extent by > grade 2 in either type or extent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2012-08; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jan Bergmanson, OD, PhD, Principal Investigator — University of Houston College of Optometry, TERTC
Locations (1):
- University of Houston College of Optometry, TERTC, Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Each subject will be randomized to wear the test lens in one eye and the control lens in the other eye. The subject is expected to attend the baseline visit not wearing their habitual contact lens products for at least 12 hours.
Groups:
- Overall Study Participants: Senofilcon A and Comfilcon A
Period: Overall Study
Arm/Group | Overall Study Participants
Started | 61
Completed | 61
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Subjects
Arm/Group | Overall Study Participants
Number analyzed (Participants) | 61
Age, Customized [Number; unit: eyes]
  <=18 years | 0
  Between 18 and 65 years | 61
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 26 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38
  Male | 23
Region of Enrollment [Number; unit: participants]
  United States | 61

OUTCOME MEASURES:

1. Primary Outcome: Subjective Responses for Comfort Rated on a 0-100 Visual Scale.
Description: Subjective Patient Ratings measured using a Visual Analog Scale on a 0-100. (0=Cannot be worn. Causes pain, 20=Frequently irritating, 40=Occasionally irritating, 60=Occasionally noticeable but not irritating, 80=Rarely noticeable, 100=Cannot be felt ever)
Time Frame: Baseline Insertion, 10 Minutes, 5 hours and 10 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Comfilcon A: comfilcon A (CooperVision Biofinity®Sphere)
- Senofilcon A: Senofilcon A (Vistakon Acuvue® Oasys)
Arm/Group | Comfilcon A | Senofilcon A
Number analyzed (Participants) | 61 | 61
units on a scale
  Baseline Insertion | 86 (15) | 87 (13)
  10 Minutes | 89 (14) | 91 (12)
  5 Hours | 83 (19) | 84 (18)
  10 Hours | 79 (23) | 81 (21)

ADVERSE EVENTS:
Groups:
- Comfilcon A: Comfilcon A / CooperVision Biofinity Sphere
Arm/Group | Overall Study Participants | Comfilcon A
Serious Adverse Events (participants affected / at risk) | 0/61 | 0/61
Other Adverse Events (participants affected / at risk) | 0/61 | 0/61

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less